CLINICAL TRIAL: NCT05483829
Title: AIDA - A Digital Health Intervention Based on Artificial Intelligence to Support the Personalized Recovery of Long COVID Patients: Feasibility Study.
Brief Title: Digital Health Intervention Based on Artificial Intelligence to Support the Personalized Recovery of Long COVID Patients Affected by Fatigue (AIDA)
Acronym: AIDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adhera Health, Inc. (Industry)
Collaborators: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FAT-22-001
Record Dates: First submitted 2022-07-28; First posted 2022-08-02 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Post Acute COVID-19 Syndrome
Keywords: Long COVID; mhealth; digital health; emotional health; behavioral intervention; mental wellbeing; mood disturbance; emotional adjustment
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Long COVID prospective group (Experimental)
  Interventions: Behavioral: Adhera® Fatigue for Long COVID program

INTERVENTIONS:
Behavioral: Adhera® Fatigue for Long COVID program — Adhera® for the Long COVID program, which includes an application and a smartwatch, supported by digital health solution based on emotional and behavioral change techniques. Patient Adaptative Self-Management Content (e.g. psycho-educational content, activities for mental wellbeing, personalized motivational messages), and the personalization is based on Adhera® Health Recommender System.
  Wearable devices and the mobile app will be used to collect real-time data for 4 weeks to detect biometric and psychometric (patient-reported outcomes) information.

SUMMARY:
The AIDA feasibility study builds upon mental health and technology acceptance theoretical frameworks. It examines the feasibility of a mobile-based digital program to support patients with long covid affected by fatigue. The program Adhera ® Fatigue Self-management is adapted for long covid patients.

DETAILED DESCRIPTION:
The study will explore the usability and engagement of a digital program designed for long covid patients affected by fatigue. The digital program relies on the Adhera® personalized digital health solution that includes personalized patient education and support, monitoring using psychometrics and wearables, and mental wellbeing exercises. The patients access the mobile solution via a mobile app. A total of 15 patients will be recruited and use the mobile solution for one month.

ELIGIBILITY:
Inclusion Criteria:

* Legal adults (older than 18)
* Long COVID diagnosis within the last year
* In possession of a compatible smartphone (Android OS v4.4 or higher)
* Reporting any of these symptoms:

  * Fatigue
  * Dyspnea
  * Anxiety
  * Stress
  * Depression
  * Sleep disorder

Exclusion Criteria:

* Hospital admission during follow-up due to pathology not related to COVID-19
* Patients without digital literacy or who cannot use the mobile application.
* Known severe psychiatric illness or cognitive impairment
* Being pregnant (or suspected to be pregnant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2022-08-28 (Actual)

PRIMARY OUTCOMES:
Behavioral outcome: Usability | At week 4
  mHealth solution usability assessed with the System Usability Scale (SUS) questionnaire. SUS can range between 0 and 100 scores, with higher values representing higher usability.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Vidal-Alaball, MD, PhD, Principal Investigator — Institut Universitari per a la recerca a l'Atencio Primaria de Salut Jordi Gol i Gurina (IDIAPJGol)
Locations (1):
- Gerencia Territorial de la Catalunya Central - Institut Catala de la Salut, Sant Fruitós de Bages, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Withings Scanwatch wearable — https://www.withings.com/de/en/scanwatch